CLINICAL TRIAL: NCT06106854
Title: Improving Medication Adherence and Outcomes in Turkish Adult Kidney Transplant Patients Using a Personal Systems Approach: SystemCHANGE™ Results of the Turkish MAGIC Randomized Clinical Trial
Brief Title: Medication Adherence in Kidney Transplant Patients: SystemCHANGE™ Results of the Turkish MAGIC Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Yaprak S. Ordin, Associate Professor Doctor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 218S720
Record Dates: First submitted 2023-09-29; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-09

CONDITIONS: Medication Adherence
Keywords: medication adherence; immunosuppressive medications; adult kidney transplant recipients; nursing; SystemCHANGE
MeSH Terms: conditions — Medication Adherence | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Behavioral: SystemCHANGE
- Control (Placebo Comparator)
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: Behavioral: SystemCHANGE — six-month SystemCHANGE™ intervention
  Arms: Intervention
Other: Education — Six patient education booklets
  Arms: Control

SUMMARY:
The SystemCHANGETM intervention harnesses patients' established daily routines/habits, environment, and important others, as possible solutions that are reoccurring and thus reliable systems that could support medication taking to become a dependable routine/habit. The aim of this study was to evaluate the effect of a six-month SystemCHANGE™ intervention compared to a six-month attention-control education intervention on medication adherence in adult kidney transplant recipients.

ELIGIBILITY:
The inclusion criteria were patients having only kidney transplantation, aged 18 years or older, taking only immunosuppressant therapy twice daily, not staying in hospital and not diagnosed with a disease shortening their life span. They also were required to own a telephone, use an electronic medication cap and bottle, understand and speak Turkish, and have approval from their nephrologist to participate in the study. They were also assessed in person for cognitive impairment using the Standardized Mini Mental Test. Those who received a 23 or higher score on the test were enrolled in the study sample.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
medication adherence | 12-months
  The six-month maintenance phase followed the intervention phase. In this phase, the patients continued to use the electronic medication monitoring cap and bottle. They were not contacted by the researcher until the completion of the six-month maintenance phase when they were contacted to return their electronic medication monitoring cap and Medication Event Monitoring System (MEMS) diary.

CONTACTS AND LOCATIONS:
Locations (1):
- Yaprak Sarıgöl Ordin, Izmir, Turkey (Türkiye)